CLINICAL TRIAL: NCT01415856
Title: A Randomized Double-Blind, Placebo-Controlled Study to Evaluate the Effect of Non-Invasive Pulsed Electromagnetic Fields (PEMF) on Postoperative Pain Following Total Knee Arthroplasty
Brief Title: Use of Pulsed Electromagnetic Fields for Postoperative Knee Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center for Joint Surgery and Sports Medicine, Maryland (Other)
Responsible Party: Ralph T. Salvagno, MD, Center for Joint Surgery and Sports Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Salvagno 20100977
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Osteoarthritis
Keywords: pulsed electromagnetic fields device; Torino II; postoperative knee pain; knee replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham Device (Torino II) (Placebo Comparator): Device is designed to appear to be giving treatment when it is not actually giving treatment. Patients will wear this for a duration of two weeks.
  Interventions: Device: Sham Device (Torino II)
- Active Device (Torino II) (Active Comparator): Device is giving treatment for 15 minutes every 2 hours for a total of two weeks.
  Interventions: Device: Active Device (Torino II)

INTERVENTIONS:
Device: Active Device (Torino II) — Device is giving treatment for 15 minutes every 2 hours for a total of two weeks.
  Arms: Active Device (Torino II)
Device: Sham Device (Torino II) — Device is designed to appear to be giving treatment when it is not actually giving treatment. Patients will wear this for a duration of two weeks.
  Arms: Sham Device (Torino II)

SUMMARY:
The purpose of this study is to determine whether the Torino II device, which emits a pulsed electromagnetic field), will help to decrease pain and swelling after knee replacement surgery, and thereby decrease the use of narcotic medications after surgery.

DETAILED DESCRIPTION:
The investigators are conducting a research study to determine if the Torino II, a pulsed electromagnetic fields (PEMF) device is helpful in reducing postoperative pain and swelling after total knee replacement surgery. Postoperative pain and swelling may cause discomfort that may directly influence functional recovery after surgery. By reducing pain and swelling immediately following surgery,the use of high doses of narcotic, NSAID, and Tyelenol pain killers can be reduced, and possibly avoided. Recovery can be maximized, as well.

The PEMF device that is being used (the Torino II) is distributed by Ivivi Health Sciences, and has been approved by the FDA for the treatment of pain and swelling following surgery. The device is non-invasive, and is fixed onto the outside of the dressing with Velcro straps. The device will give off electromagnetic pulses to target pain relief in the knee. PEMF devices have been in clinical use for decades, and to date, no reported side effects have occurred.

It is important to note that treatment will still follow the standard Meritus Medical Center protocol for knee replacement surgery. This includes pain medication, icing, and physical therapy. This standard protocol will be followed no matter what study group patients are assigned to. Participation in this study or lack thereof will not change the treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age: greater than 18 years
* Weight: less than 300 lbs.
* Diagnosis: osteoarthritis
* Type of Surgery: unilateral knee replacement

Exclusion Criteria:

* No pacemaker or defibrillator.
* No infection of the affected knee.
* No previous open surgery of the affected knee.
* No history of Rheumatoid Arthritis.
* No more than 2 narcotic pills per month in the last 6 months for pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Pain | 2 weeks
  Pain is measured on a scale of 0-10, which is the VAS scale used by most hospitals, including Meritus Medical Center. 0 indicates no pain, while 10 indicates the worst pain possible.
Edema (Swelling) | 2 weeks
  Swelling will be measured by using a disposable tape measure to measure the circumference of the patient's knee at the mid-patellar region. This will be measured in millimeters.

SECONDARY OUTCOMES:
Narcotic Pain Medications | 2 weeks
  Patients will record their use of pain and anti-inflammatory medications.
Range of Motion | 2 weeks
  Patient range of motion in degrees will be measured, for flexion and extension.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Joint Surgery and Sports Medicine, Hagerstown, Maryland, United States